CLINICAL TRIAL: NCT02264990
Title: A Randomized, Open-Label, Multicenter, Phase 3 Trial Comparing Veliparib Plus Carboplatin and Paclitaxel Versus Investigator's Choice of Standard Chemotherapy in Subjects Receiving First Cytotoxic Chemotherapy for Metastatic or Advanced Non-Squamous Non-Small Cell Lung Cancer (NSCLC) and Who Are Current or Former Smokers
Brief Title: Study Comparing Veliparib Plus Carboplatin and Paclitaxel Versus Investigator's Choice of Standard Chemotherapy in Adults Receiving First Cytotoxic Chemotherapy for Metastatic or Advanced Non-Squamous Non-Small Cell Lung Cancer (NSCLC) and Who Are Current or Former Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-359; 2014-002565-30 (EudraCT Number)
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: veliparib; carboplatin; paclitaxel; cisplatin; pemetrexed; Poly Adenosine diphosphate (ADP)-ribose Polymerase (PARP); Metastatic; Non-squamous; Non-small cell lung cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Cisplatin; veliparib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veliparib + Carboplatin + Paclitaxel (Experimental): Participants received 120 mg veliparib twice a day (BID) on Days -2 to 5 (7 days), carboplatin at an area under the curve (AUC) of 6 mg/mL*min on Day 1 and paclitaxel 200 mg/m² on Day 1 of each 21-day cycle for a maximum of 6 cycles.
  After completion of up to 6 cycles, optional maintenance pemetrexed was administered as 500 mg/m² on Day 1 of each 21-day cycle until toxicity required cessation of therapy, or radiographic progression occurred.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Veliparib; Drug: Pemetrexed
- Investigator's Choice Chemotherapy (Active Comparator): Participants received Investigator's choice of standard doublet chemotherapy consisting of 1 of the following 3 options, administered on Day 1 of each 21-day cycle for a maximum of 6 cycles:
  * Carboplatin AUC 6 mg/mL*min + paclitaxel 200 mg/m²
  * Cisplatin 75 mg/m² + pemetrexed 500 mg/m²
  * Carboplatin AUC 6 or AUC 5 mg/mL*min + pemetrexed 500 mg/m²
  After completion of up to 6 cycles, optional maintenance pemetrexed was administered as 500 mg/m² on Day 1 of each 21-day cycle until toxicity required cessation of therapy, or radiographic progression occurred.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Paclitaxel — Administered by Intravenous infusion on Day 1 of each 21-day cycle
Drug: Carboplatin — Administered by Intravenous infusion on Day 1 of each 21-day cycle
Drug: Cisplatin — Administered by Intravenous infusion on Day 1 of each 21-day cycle
  Arms: Investigator's Choice Chemotherapy
Drug: Veliparib — Oral capsule, administered twice daily for 7 days in each 21-day cycle
  Other Names: ABT-888
  Arms: Veliparib + Carboplatin + Paclitaxel
Drug: Pemetrexed — Administered by Intravenous infusion on Day 1 of each 21-day cycle
  Other Names: Alimta

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of veliparib plus carboplatin and paclitaxel versus the Investigator's choice of standard chemotherapy in adults with metastatic or advanced non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age with life expectancy > 12 weeks.
* Subject must have cytologically or histologically confirmed advanced or metastatic non-squamous NSCLC and are current or former smokers.
* Subject must have NSCLC that is not amenable to surgical resection or radiation with curative intent at time of screening.
* Subject must have at least 1 unidimensional measurable NSCLC lesion on a computed tomography (CT) scan as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Exclusion Criteria:

* Subject has a known hypersensitivity to paclitaxel or to other drugs formulated with polyethoxylated castor oil (Cremophor).
* Subject has a known hypersensitivity to platinum compounds.
* Subject has peripheral neuropathy ≥ grade 2.
* Subject has squamous NSCLC, or an untreated known epidermal growth factor receptor (EGFR) mutation of exon 19 deletion or L858R mutation in exon 21, or a known anaplastic lymphoma kinase (ALK) gene rearrangement.
* Subject has received prior cytotoxic chemotherapy or chemoradiotherapy for NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (140):
- United States (25):
  - Clearview Cancer Institute /ID# 131434, Huntsville, Alabama
  - University of South Alabama /ID# 131518, Mobile, Alabama
  - Highlands Oncology Group /ID# 131250, Springdale, Arkansas
  - CBCC Global Research, Inc. at /ID# 132709, Bakersfield, California
  - California Cancer Assoc. R&E /ID# 131392, Encinitas, California
  - California Cancer Assoc. R&E /ID# 131949, Encinitas, California
  - LA Hem-Oncology Med Group /ID# 131639, Los Angeles, California
  - St Jude Hospital dba St Joseph /ID# 132943, Santa Rosa, California
  - Icri /Id# 132942, Whittier, California
  - University of Florida - Archer /ID# 132408, Gainesville, Florida
  - NorthShore University HealthSystem - Evanston Hospital /ID# 130200, Evanston, Illinois
  - Goshen Center for Cancer Care /ID# 130216, Goshen, Indiana
  - University of Louisville /ID# 130217, Louisville, Kentucky
  - Cancer Center of Acadiana /ID# 133611, Lafayette, Louisiana
  - Henry Ford Health System /ID# 130234, Detroit, Michigan
  - Herbert Herman Cancer Center /ID# 130239, Lansing, Michigan
  - Washington University-School of Medicine /ID# 131651, St Louis, Missouri
  - MD Anderson Cancer Center at Cooper - Camden /ID# 131490, Camden, New Jersey
  - Gabrail Cancer Center Research /ID# 130205, Canton, Ohio
  - Univ Oklahoma HSC /ID# 132888, Oklahoma City, Oklahoma
  - Albert Einstein Medical Center /ID# 134498, Philadelphia, Pennsylvania
  - Allegheny General Hospital /ID# 134049, Pittsburgh, Pennsylvania
  - The Jones Clinic, PC /ID# 130215, Germantown, Tennessee
  - UT Southwestern Medical Center /ID# 130236, Dallas, Texas
  - Univ Texas HSC San Antonio /ID# 132972, San Antonio, Texas
- Argentina (4):
  - Coiba /Id# 132153, Berazategui, Buenos Aires
  - Centro Investigacion Pergamino /ID# 132152, Pergamino
  - Hospital Britanico /ID# 134874, Rosario, Santa FE
  - Instituto de Oncologia de Rosa /ID# 132150, Rosario, Santa FE
- Australia (4):
  - St George Hospital /ID# 132481, Kogarah, New South Wales
  - Southern Medical Day Care Ctr /ID# 132482, Wollongong, New South Wales
  - Flinders Centre for Innovation /ID# 134288, Bedford Park, South Australia
  - Royal Hobart Hospital /ID# 132477, Hobart, Tasmania
- Canada (4):
  - Qe Ii Hsc /Id# 133408, Halifax, Nova Scotia
  - Victoria Hospital /ID# 132161, London, Ontario
  - Windsor Regional Hospital /ID# 135989, Windsor, Ontario
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 132155, Québec, Quebec
- Czechia (4):
  - Krajska nemocnice Liberec a.s. /ID# 132694, Liberec
  - Univ Hosp Ostrava-Poruba /ID# 132690, Ostrava
  - Multiscan s.r.o. /ID# 132689, Pardubice
  - Vseobecna Fakultni Nemocnice /ID# 135118, Prague
- Odense Universitets Hospital /ID# 131912, Odense C, Region Syddanmark, Denmark
- Finland (2):
  - Satakunnan Sairaanhoitopiiri /ID# 133632, Pori
  - Vaasa Central Hospital /ID# 131930, Vaasa
- Germany (4):
  - Charite-Univ. Berlin, Benjamin-Franklin /ID# 131927, Berlin
  - Lungen Clinic Grosshansdorf /ID# 131928, Großhansdorf
  - Univ Klinik Eppendorf Hamburg /ID# 131926, Hamburg
  - Klinik Loewenstein GmbH /ID# 131925, Löwenstein
- Hungary (7):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 133441, Miskolc, Borsod-Abauj Zemplen county
  - Orszagos Koranyi Pulmonologiai Intezet /ID# 132738, Budapest XII, Budapest
  - Debreceni Egyetem Klinikai Kozpont /ID# 132742, Debrecen
  - Koch Robert Hospital /ID# 133440, Edelény
  - Veszprem Megyei Tudogyogyintez /ID# 132739, Farkasgyepű
  - Petz Aladar Megyei Oktato Korh /ID# 132741, Győr
  - Matrahaza Gyogyintezet /ID# 132743, Kékesteto
- Israel (4):
  - Assaf Harofeh Medical Center /ID# 132830, Be’er Ya‘aqov
  - Shaare Zedek Medical Center /ID# 132834, Jerusalem
  - Meir Medical Center /ID# 132832, Kfar Saba
  - Sheba Medical Center /ID# 132833, Ramat Gan
- Japan (12):
  - Aichi Cancer Center Hospital /ID# 134129, Nagoya, Aichi-ken
  - Kurume University Hospital /ID# 134117, Kurume-shi, Fukuoka
  - Hokkaido University Hospital /ID# 134123, Sapporo, Hokkaido
  - Kanagawa Cardiovascular and Respiratory Center /ID# 134127, Yokohama, Kanagawa
  - Sendai Kousei Hospital /ID# 135491, Sendai, Miyagi
  - Osaka City General Hospital /ID# 134115, Osaka, Osaka
  - Kindai University Hospital /ID# 134112, Osaka-sayama-shi, Osaka
  - National Cancer Center Hospital /ID# 135129, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 135492, Koto-ku, Tokyo
  - Yamaguchi - Ube Medical Center /ID# 135284, Ube-shi, Yamaguchi
  - Hiroshima Citizens Hospital /ID# 135130, Hiroshima
  - Kishiwada City Hospital /ID# 136548, Kishiwada
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis /ID# 131968, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum /ID# 131967, Amsterdam
  - Catharina Ziekenhuis /ID# 131966, Eindhoven
  - Ziekenhuis St. Jansdal /ID# 131965, Harderwijk
  - St. Antonius Ziekenhuis /ID# 133635, Nieuwegein
- New Zealand (2):
  - Canterbury District Health Boa /ID# 132469, Christchurch
  - Wellington Hospital (Capital and Coast District Health Board) /ID# 132470, Wellington
- Russia (12):
  - Federal State Budgetary Scientific Institution N.N. Blokhin Russian Cancer Resea /ID# 137085, Moscow, Moscow
  - Sverdlovsk Regional Oncology Center Dispensary /ID# 132375, Yekaterinburg, Sverdlovsk Oblast
  - archangel Clinical Oncology /ID# 132376, Arkhangelsk
  - Moscow Regional Onc Dispensary /ID# 132381, Balashikha
  - Belgorod Oncology Dispensary /ID# 142638, Belgorod
  - Moscow Res Onc Inst Hertsen /ID# 132370, Moscow
  - State Regional Budgetary Healthcare Institution " Murmansk Regional Oncology Dis /ID# 137087, Murmansk
  - Orenburg Regional Clinical Onc /ID# 132371, Orenburg
  - Strategic medical systems LLC /ID# 206383, Saint Petersburg
  - LLC BioEq Ltd. /ID# 132372, Saint Petersburg
  - N.N. Petrov Research Inst Onc /ID# 137084, Saint Petersburg
  - Ogarev Mordovia State Univ /ID# 132377, Saransk
- South Africa (8):
  - GVI Oncology /ID# 133268, Port Elizabeth, Eastern Cape
  - Dr Albert, Bouwer and Jordaan Incorporated /ID# 131775, Pretoria, Gauteng
  - Mary Potter Oncology Centre /ID# 131776, Pretoria, Gauteng
  - The Oncology Centre /ID# 131773, Durban, KwaZulu-Natal
  - Netcare Oncology Intervent Ctr /ID# 131777, Cape Town, Western Cape
  - Cape Town Oncology Trials /ID# 132734, Cape Town, Western Cape
  - GVI Rondebosch Oncology Centre /ID# 132732, Cape Town, Western Cape
  - Sandton Oncology Medical Group /ID# 131774, Johannesburg
- South Korea (6):
  - Dong-A University Hospital /ID# 131609, Busan, Busan Gwang Yeogsi
  - Seoul National Univ Bundang ho /ID# 131610, Seongnam, Gyeonggido
  - Inha University Hospital /ID# 147924, Junggu, Incheon Gwang Yeogsi
  - Chonnam National University Hospital /ID# 131612, Gwangju, Jeonranamdo
  - Samsung Medical Center /ID# 132471, Seoul, Seoul Teugbyeolsi
  - Chungbuk National Univ Hosp /ID# 131611, Cheongju-si
- Spain (9):
  - Hospital Duran i Reynals /ID# 132879, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Fundacion Alcorcon /ID# 132909, Alcorcón
  - Hospital General Universitario Alicante /ID# 132881, Alicante
  - Hospital Universitario Dexeus - Grupo Quironsalud /ID# 132876, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 132871, Barcelona
  - MD Anderson Madrid /ID# 132905, Madrid
  - Hospital Universitario La Paz /ID# 132870, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 132869, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 132873, Valencia
- Taiwan (4):
  - China Medical University Hosp /ID# 131870, Taichung, Taichung
  - Dalin Tzu Chi General Hospital /ID# 131872, Dalin Township
  - Taipei Medical University Hospital /ID# 133817, Taipei
  - Taipei Veterans General Hosp /ID# 131871, Taipei
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty /ID# 131913, Ankara
  - Ankara Univ Medical Faculty /ID# 131914, Ankara
  - Uludag University Medical Faculty /ID# 131915, Bursa
  - Dicle Universitesi Tip /ID# 136570, Diyarbakır
  - Gaziantep Universitesi Med /ID# 131917, Gaziantep
  - Dr. Suat Seren Gogus Has /ID# 136568, Izmir
  - Inonu University /ID# 136569, Malatya
- United Kingdom (16):
  - Leicester Royal Infirmary /ID# 133930, Leicester, England
  - Cheltenham General Hospital /ID# 131951, Cheltenham, Gloucestershire
  - Norfolk and Norwich Univ Hosp /ID# 131953, Norwich, Norfolk
  - Royal United Hospitals Bath /ID# 132851, Bath
  - Belfast City Hospital /ID# 132858, Belfast
  - Heart of England NHS Foundation Trust /ID# 132855, Birmingham
  - Royal Blackburn Hospital /ID# 132853, Blackburn
  - Colchester General Hospital /ID# 133929, Colchester
  - Castle Hill Hospital /ID# 135489, Cottingham
  - Scunthorpe General Hospital /ID# 133931, Doncaster
  - James Paget University Hosp /ID# 131954, Great Yarmouth
  - Royal Gwent Hospital /ID# 133935, Gwent
  - Huddersfield Royal Infirmary /ID# 132854, Huddersfield
  - Charing Cross Hospital /ID# 131959, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust Freeman Hospital /ID# 131661, Newcastle upon Tyne
  - York Hospital /ID# 132859, York

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Govindan R, Lind M, Insa A, Khan SA, Uskov D, Tafreshi A, Guclu S, Bar J, Kato T, Lee KH, Nakagawa K, Hansen O, Biesma B, Kundu MG, Dunbar M, He L, Ansell P, Sehgal V, Huang X, Glasgow J, Bach BA. Veliparib Plus Carboplatin and Paclitaxel Versus Investigator's Choice of Standard Chemotherapy in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer. Clin Lung Cancer. 2022 May;23(3):214-225. doi: 10.1016/j.cllc.2022.01.005. Epub 2022 Feb 4. PMID 35331641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 131 sites in 20 countries (Argentina, Australia, Canada, Czech Republic, Denmark, Finland, Germany, Hungary, Israel, Japan, South Korea, Netherlands, New Zealand, Russian Federation, South Africa, Spain, Taiwan, Turkey, United Kingdom, and United States).
Pre-assignment Details: Participants were randomized in a 1:1 ratio to veliparib in combination with carboplatin and paclitaxel (C/P) or investigator's choice of platinum doublet chemotherapy. Randomization was stratified by smoking status (current versus former), by the investigators' preferred platinum doublet therapy (carboplatin/paclitaxel versus cisplatin/pemetrexed versus carboplatin/pemetrexed), by gender (male versus female) and by Eastern Cooperative Oncology Group (ECOG) performance status (0 versus 1).
Groups:
- Investigator's Choice Chemotherapy: Participants received investigator's choice of standard doublet chemotherapy consisting of 1 of the following 3 options, administered on Day 1 of each 21-day cycle for a maximum of 6 cycles:
  * Carboplatin at an area under the curve (AUC) of 6 mg/mL*min + paclitaxel 200 mg/m²
  * Cisplatin 75 mg/m² + pemetrexed 500 mg/m²
  * Carboplatin AUC 6 or AUC 5 mg/mL*min + pemetrexed 500 mg/m²
  After completion of up to 6 cycles, optional maintenance pemetrexed was administered as 500 mg/m² on Day 1 of each 21-day cycle until toxicity required cessation of therapy, or radiographic progression occurred.
- Veliparib + Carboplatin + Paclitaxel: Participants received 120 mg veliparib twice a day (BID) on Days -2 to 5 (7 days), carboplatin at an AUC of 6 mg/mL*min on Day 1 and paclitaxel 200 mg/m² on Day 1 of each 21-day cycle for a maximum of 6 cycles.
  After completion of up to 6 cycles, optional maintenance pemetrexed was administered as 500 mg/m² on Day 1 of each 21-day cycle until toxicity required cessation of therapy, or radiographic progression occurred.
Period: Overall Study
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Started | 297 | 298
Received Treatment | 288 | 293
Received Maintenance Therapy | 148 | 123
Completed | 37 | 39
Not Completed | 260 | 259
Not completed — Death | 255 | 250
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all randomized participants.
Groups:
- Veliparib + Carboplatin + Paclitaxel: Participants received 120 mg veliparib BID on Days -2 to 5 (7 days), carboplatin at an AUC of 6 mg/mL*min on Day 1 and paclitaxel 200 mg/m² on Day 1 of each 21-day cycle for a maximum of 6 cycles.
  After completion of up to 6 cycles, optional maintenance pemetrexed was administered as 500 mg/m² on Day 1 of each 21-day cycle until toxicity required cessation of therapy, or radiographic progression occurred.
- Total: Total of all reporting groups
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel | Total
Number analyzed (Participants) | 297 | 298 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.99) | 62.7 (9.02) | 62.9 (9.0)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 153 | 163 | 316
  ≥ 65 years | 144 | 135 | 279
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 92 | 182
  Male | 207 | 206 | 413
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 26 | 48
  Not Hispanic or Latino | 275 | 272 | 547
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 233 | 229 | 462
  Black | 11 | 11 | 22
  Asian | 53 | 57 | 110
  Other | 0 | 1 | 1
Region [Count of Participants; unit: Participants]
  US and Western Europe and Australia and Canada | 177 | 157 | 334
  Eastern Europe/Russia | 68 | 88 | 156
  Japan | 37 | 35 | 72
  Other Asian | 15 | 18 | 33
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 153 | 152 | 305
  Past smoker | 144 | 146 | 290
Investigators' Preferred Platinum Doublet Therapy [Count of Participants; unit: Participants] — The investigator's preferred choice of platinum doublet therapy, prior to randomization, which was used as a stratification factor. Note that while the investigator's pre-randomization preferred choice for the doublet is summarized, all participants on the veliparib arm received carboplatin and paclitaxel as chemotherapy.
  Participants
    Carboplatin/paclitaxel | 71 | 70 | 141
    Cisplatin/pemetrexed | 95 | 100 | 195
    Carboplatin/pemetrexed | 131 | 128 | 259
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  * 0 = Fully Active;
  * 1 = Restricted activity but ambulatory;
  * 2 = Ambulatory but unable to carry out work activities;
  * 3 = Limited Self-Care;
  * 4 = Completely Disabled, No self-care
  Participants
    Grade 0 (fully active) | 113 | 116 | 229
    Grade 1 (restricted but ambulatory) | 184 | 182 | 366
Lung Subtype Panel (LSP) Assay Results [Count of Participants; unit: Participants] — LSP positive: Patients with tumors classified as positive for the gene expression-based lung subtype panel (LSP) biomarker
  LSP negative: Patients with tumors classified as negative for the gene expression-based lung subtype panel (LSP) biomarker Population: Participants with a tumor tissue sample available with sufficient tumor content for LSP status evaluation, and with an analytically valid LSP result.
  Participants
    number analyzed (Participants) | 93 | 114 | 207
    LSP positive | 40 | 40 | 80
    LSP negative | 53 | 74 | 127

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the Lung Subtype Panel Positive Subgroup
Description: Overall survival is defined as the time from the date that the participant was randomized to the date of the participant's death. Overall survival was estimated using Kaplan-Meier methodology. Participants still alive at the data cut-off date were censored at the date they were last known to be alive.
Time Frame: From randomization up to the data cut-off date of 15 July 2019; median follow-up time was 44.5 and 45.3 months in LSP+ participants for the investigator's choice chemotherapy and veliparib + C/P arms, respectively.
Population: Participants in the ITT population who were LSP positive (LSP+)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Number analyzed (Participants) | 40 | 40
months | 9.2 [5.1 to 11.7] | 11.2 [7.5 to 15.8]
Statistical Analysis 1: Comparison: Investigator's Choice Chemotherapy vs Veliparib + Carboplatin + Paclitaxel; Test type: Superiority — A fixed sequence testing procedure was used for analyses of the primary and secondary efficacy endpoints to control for the familywise error rate. If veliparib plus C/P treatment was not statistically significantly better compared to the investigators' choice of standard therapy for the primary efficacy endpoint of OS in LSP+ participants, then statistical significance would not be declared for any of the secondary efficacy endpoints; p = 0.113, Log Rank — Statistical significance was determined by a two-sided P value ≤ 0.05; Log rank test stratified by ECOG performance status, investigators' preferred platinum therapy, and gender; Hazard Ratio (HR) = 0.644, 95% CI 2-sided [0.396 to 1.048] — Hazard ratio obtained using the covariate adjusted Cox Proportional Hazard Model with covariates being ECOG performance status, investigators' preferred platinum therapy, and gender

2. Secondary Outcome: Progression Free Survival (PFS) in the Lung Subtype Panel Positive Subgroup
Description: Progression-free survival is defined as the time from the date of randomization to the date of disease progression (PD) per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or death (all causes of mortality), whichever occurred first.
  PD: At least a 20% increase in the size of target lesions, taking as reference the smallest size recorded since the treatment started (Baseline or after) with an absolute increase of at least 5 mm, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
  PFS was estimated using Kaplan-Meier methodology. Participants who did not have an event of disease progression or had not died on or before the cutoff date were censored at the date of their last disease progression assessment on or before the cut-off date. Any PD and death occurring > 26 weeks and > 12 weeks after the previous assessment, respectively, were excluded and patients were censored at last assessment before PD or death.
Time Frame: From randomization up to the data cut-off date of 15 July 2019; the median follow-up time was 44.5 and 45.3 months in LSP+ participants for the investigator's choice chemotherapy and veliparib + C/P arms, respectively.
Population: Participants in the ITT population who were LSP positive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Number analyzed (Participants) | 40 | 40
months | 5.2 [2.8 to 6.2] | 6.3 [3.5 to 7.4]
Statistical Analysis 1: Comparison: Investigator's Choice Chemotherapy vs Veliparib + Carboplatin + Paclitaxel; Test type: Other; p = 0.260, Log Rank; Log-rank test stratified by investigator's preferred platinum therapy, gender, and ECOG performance status; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.388 to 1.080] — The hazard ratio was obtained using the covariate adjusted Cox Proportional Hazard Model with covariates of ECOG performance status, investigators' preferred platinum therapy, and gender

3. Secondary Outcome: Objective Response Rate (ORR) in the Lung Subtype Panel Positive Subgroup
Description: Objective response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria. Response must have been confirmed at a consecutive assessment 28 days or more after the assessment at which response was first observed.
  CR: The disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters, persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, or any new lesions.
Time Frame: Assessed on Day 1 of Cycles 3 and 5 then every 9 weeks for 1 year or until maintenance therapy was discontinued, then every 12 weeks until radiographic progression or death; median time on follow-up was 5.2 and 6.3 months in each group, respectively.
Population: Participants in the ITT population who were LSP positive
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Number analyzed (Participants) | 40 | 40
percentage of participants | 30.0 [16.6 to 46.5] | 22.5 [10.8 to 38.5]
Statistical Analysis 1: Comparison: Investigator's Choice Chemotherapy vs Veliparib + Carboplatin + Paclitaxel; Test type: Other; p = 0.455, Regression, Logistic; Logistic regression adjusted for the covariates of ECOG performance status, investigators' preferred platinum therapy, and gender; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.23 to 1.90] — Odds ratio is from covariate adjusted logistic regression with the covariates being ECOG performance status, investigators' preferred platinum therapy, and gender

4. Secondary Outcome: Overall Survival in All Participants
Description: Overall survival is defined as the time from the date that the participant was randomized to the date of the participant's death. OS was estimated using Kaplan-Meier methodology. Participants still alive at the data cut-off date were censored at the date they were last known to be alive.
Time Frame: From randomization up to the data cut-off date of 15 July 2019; the median OS follow-up time was 45.4 and 44.6 months in all participants for the investigator's choice chemotherapy and veliparib + C/P arms, respectively.
Population: Participants in the ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Number analyzed (Participants) | 297 | 298
months | 12.1 [10.0 to 13.7] | 12.1 [10.4 to 14.9]
Statistical Analysis 1: Comparison: Investigator's Choice Chemotherapy vs Veliparib + Carboplatin + Paclitaxel; Test type: Other; p = 0.846, Log Rank; Log rank test stratified by LSP status, ECOG performance status, investigators' preferred platinum therapy, and gender; Hazard Ratio (HR) = 0.986, 95% CI 2-sided [0.827 to 1.176] — The hazard ratio was obtained using the covariate adjusted Cox Proportional Hazard Model with covariates of LSP status, ECOG performance status, investigators' preferred platinum therapy, and gender

5. Secondary Outcome: Progression Free Survival (PFS) in All Participants
Description: Progression-free survival is defined as the time from the date of randomization to the date of disease progression (PD) per RECIST version 1.1 or death (all causes of mortality), whichever occurred first.
  PD: At least a 20% increase in the size of target lesions, taking as reference the smallest size recorded since the treatment started (Baseline or after) with an absolute increase of at least 5 mm, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
  PFS was estimated using Kaplan-Meier methodology. Participants who did not have an event of disease progression or had not died on or before the cut-off date were censored at the date of their last disease progression assessment on or before the cut-off date. Any PD and death occurring > 26 weeks and > 12 weeks after the previous assessment, respectively, were excluded and patients were censored at last assessment before PD or death.
Time Frame: From randomization up to the data cut-off date of 15 July 2019; the median follow-up time was 45.4 and 44.6 months in all participants for the investigator's choice chemotherapy and veliparib + C/P arms, respectively.
Population: Participants in the ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Number analyzed (Participants) | 297 | 298
months | 6.7 [5.6 to 7.2] | 5.9 [5.0 to 6.5]
Statistical Analysis 1: Comparison: Investigator's Choice Chemotherapy vs Veliparib + Carboplatin + Paclitaxel; Test type: Other; p = 0.473, Log Rank; Log rank test stratified by LSP status, ECOG performance status, investigators' preferred platinum therapy, and gender; Hazard Ratio (HR) = 1.035, 95% CI 2-sided [0.867 to 1.235] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Objective Response Rate (ORR) in All Participants
Description: Objective response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) per RECIST version 1.1 criteria. Response must have been confirmed at a consecutive assessment 28 days or more after the assessment at which response was first observed.
  CR: The disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters, persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, or any new lesions.
Time Frame: Assessed on Day 1 of Cycles 3 and 5 then every 9 weeks for 1 year or until maintenance therapy was discontinued, then every 12 weeks until radiographic progression or death; median time on follow-up was 6.7 and 5.9 months in each group, respectively.
Population: Participants in the ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
Number analyzed (Participants) | 297 | 298
percentage of participants | 29.0 [23.9 to 34.5] | 26.2 [21.3 to 31.6]
Statistical Analysis 1: Comparison: Investigator's Choice Chemotherapy vs Veliparib + Carboplatin + Paclitaxel; Test type: Other; p = 0.409, Regression, Logistic; Logistic regression adjusted for the covariates of LSP status, ECOG performance status, investigators' preferred platinum therapy, and gender; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.59 to 1.24] — Odds ratio is from covariate adjusted logistic regression with the covariates being LSP status, ECOG performance status, investigators' preferred platinum therapy, and gender

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization until the end of study; the median follow-up time was 45.4 and 44.6 months in each treatment group, respectively. Adverse events: From first dose of study drug until 30 days after last dose of study drug (veliparib or investigators' choice of standard chemotherapy); median duration of treatment ranged from 86 to 111 days for each treatment.
Description: All-cause mortality is reported for all randomized participants. Adverse events are reported for the as-treated subjects population, which included all participants who received at least 1 dose of study drug (veliparib/investigator's choice of standard chemotherapy).
Arm/Group | Investigator's Choice Chemotherapy | Veliparib + Carboplatin + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 255/297 | 250/298
Serious Adverse Events (participants affected / at risk) | 98/288 | 121/293
Other Adverse Events (participants affected / at risk) | 269/288 | 275/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigator's Choice Chemotherapy (N=288) | Veliparib + Carboplatin + Paclitaxel (N=293)
ANAEMIA (Blood and lymphatic system disorders) | 15 (17) | 7 (8)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7 (10) | 13 (15)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 6 (9)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 4 (4)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 2 (2)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 7 (7)
PERICARDITIS (Cardiac disorders) | 1 (2) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (4) | 2 (2)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 5 (5) | 6 (6)
ASTHENIA (General disorders) | 2 (2) | 1 (2)
CATHETER SITE HAEMORRHAGE (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 2 (2) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (2) | 0 (0)
MALAISE (General disorders) | 3 (6) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 2 (2) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (2)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0)
SUDDEN DEATH (General disorders) | 1 (1) | 2 (2)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 3 (4)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 (0) | 1 (1)
EMPYEMA (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 2 (2) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 4 (4)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (2)
LYMPHANGITIS (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 8 (9) | 19 (26)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
SEPSIS (Infections and infestations) | 4 (5) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEART INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (12) | 14 (19)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 2 (2)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (1)
AZOTAEMIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (8)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 5 (7)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ANEURYSM (Vascular disorders) | 0 (0) | 1 (1)
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 2 (2)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigator's Choice Chemotherapy (N=288) | Veliparib + Carboplatin + Paclitaxel (N=293)
ANAEMIA (Blood and lymphatic system disorders) | 107 (197) | 112 (212)
LEUKOPENIA (Blood and lymphatic system disorders) | 40 (77) | 43 (77)
NEUTROPENIA (Blood and lymphatic system disorders) | 89 (175) | 104 (210)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 54 (102) | 76 (155)
CONSTIPATION (Gastrointestinal disorders) | 92 (113) | 69 (81)
DIARRHOEA (Gastrointestinal disorders) | 47 (60) | 51 (70)
NAUSEA (Gastrointestinal disorders) | 131 (202) | 86 (121)
STOMATITIS (Gastrointestinal disorders) | 30 (32) | 19 (24)
VOMITING (Gastrointestinal disorders) | 73 (99) | 39 (48)
ASTHENIA (General disorders) | 30 (50) | 29 (58)
FATIGUE (General disorders) | 89 (117) | 80 (108)
OEDEMA PERIPHERAL (General disorders) | 24 (36) | 13 (16)
PYREXIA (General disorders) | 16 (21) | 15 (17)
WEIGHT DECREASED (Investigations) | 24 (25) | 14 (17)
DECREASED APPETITE (Metabolism and nutrition disorders) | 79 (109) | 63 (79)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 11 (15) | 24 (24)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 16 (19) | 21 (22)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 12 (14) | 16 (18)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 26 (35) | 39 (45)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 22 (24) | 17 (21)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 9 (13) | 15 (21)
MYALGIA (Musculoskeletal and connective tissue disorders) | 17 (22) | 38 (50)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 15 (19) | 15 (17)
DIZZINESS (Nervous system disorders) | 22 (25) | 17 (17)
DYSGEUSIA (Nervous system disorders) | 29 (33) | 19 (20)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 42 (51) | 131 (195)
INSOMNIA (Psychiatric disorders) | 30 (30) | 37 (39)
COUGH (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 27 (32)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 25 (30) | 42 (46)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 21 (29) | 17 (27)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 6 (8)
ALOPECIA (Skin and subcutaneous tissue disorders) | 34 (40) | 137 (160)
RASH (Skin and subcutaneous tissue disorders) | 25 (29) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02264990/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02264990/SAP_001.pdf